CLINICAL TRIAL: NCT05391867
Title: Assessment of the Efficacy of Lenvatinib Versus Sorafenib in the Management of Advanced Hepatocellular Carcinoma - An Open-label Randomized Clinical Control Trial in a Tertiary Care Hospital.
Brief Title: Assessment of the Efficacy of Lenvatinib Versus Sorafenib in the Management of Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Salimullah Medical College Mitford Hospital (Other Government)
Responsible Party: Principal Investigator, Md. Fazal Karim, Associate Professor, Sir Salimullah Medical College Mitford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sirsalimullah
Record Dates: First submitted 2020-11-26; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Sorafenib

STUDY DESIGN:
Intervention Model Description: An open label randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenvatinib group (Group-A) (Experimental): Patients diagnosed as hepatocellular carcinoma will be randomly assigned for treatment with Lenvatinib. Cap. Lenvatinib will be given at doses of 4 mg 12 hourly.
  Interventions: Drug: Lenvatinib
- Sorafenib group (Group-B) (Experimental): Patients diagnosed as hepatocellular carcinoma will be randomly assigned for treatment with Sorafenib. Tab. Sorafenib will be given at doses of 200 mg 12 hourly.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Tyrosine kinase inhibitor
  Other Names: Sorafenib

SUMMARY:
Hepatocellular carcinoma is the most common type of liver cancer, which is the 3rd leading cause of cancer deaths worldwide. The incidence is expected to increase as a consequence of chronic liver disease with its multiple risk factors, including chronic hepatitis B virus (HBV) and hepatitis C virus (HCV) infections, excessive alcohol consumption, nonalcoholic fatty liver disease, hemochromatosis, and aflatoxin B1.It is estimated that 70%-90% of patients with HCC have chronic liver disease and cirrhosis, which limits the feasibility of surgical procedures in advanced cases. There are limited treatment options for HCC patients who are ineligible for surgical resection. Locoregional therapies, such as radiofrequency ablation, transarterial chemoembolization (TACE), transarterial embolization (TAE), or hepatic arterial infusion chemotherapy (HAIC), are primarily recommended, and if one of those fail, then systemic therapy is considered. The 2013 Japan Society of Hepatology HCC Guidelines outlined that the factors influencing treatment decisions should be based on the degree of liver damage (Child-Pugh), presence or absence of extrahepatic spread and macrovascular invasion, the number of tumors, and tumor diameter. Sorafenib has been the standard of care since 2007, when the SHARP trial demonstrated that sorafenib improved median overall survival (OS) compared to placebo in patients who had not received prior systemic therapy (10.7 vs 7.9 months, HR =0.69, P<0.001). In patients from the Asia-Pacific region taking sorafenib, the median improvement in overall survival compared with placebo was 2.3 months (6.5 months vs 4.2 months; HR 0.68; p=0.014). Drug development for hepatocellular carcinoma in the past 10 years has been marked by four failed global phase 3 trials (of sunitinib, brivanib, linifanib, and erlotinib plus sorafenib) that did not show non-inferiority. Sorafenib, an oral multikinase inhibitor, has been the only systemic therapy demonstrated to extend overall survibility as a firstline treatment, showing a median improvement of 2.8 months compared with placebo (10.7 months vs. 7.9 months; hazard ratio [HR] 0.69; p\0.001).6 Inpatients from the Asia-Pacific region taking sorafenib, the median OS (mOS) improvement compared with placebo was 2.3 months (HR 0.68; p = 0.014). The use of other molecularly targeted agents has not demonstrated efficacy via non-inferiority or superiority to sorafenib; thus, until the appearance of lenvatinib, sorafenib has also been widely used as the first-line treatment for uHCC patients in Japan. Recently, regorafenib and Nivolumab were approved as a second-line systemic treatment for patients who do not respond to the first-line treatments. Otherwise, best supportive care or participation in clinical trials is recommended in the second-line setting by treatment guidelines. Chemotherapy in combination with sorafenib (doxorubicin) and radioembolization with SIR Spheres Y-90 resin microspheres failed to demonstrate a survival benefit or showed a worse safety profile compared to sorafenib in the first-line setting. Eventually, the PhaseIII non-inferiority REFLECT trial showed that lenvatinib was non-inferior compared to sorafenib.

DETAILED DESCRIPTION:
1. Introduction:

   Hepatocellular carcinoma is one of the most common type of liver cancer, which is the 3rd leading cause of cancer deaths worldwide. The incidence is expected to increase as a consequence of chronic liver disease with its multiple risk factors, including chronic hepatitis B virus (HBV) and hepatitis C virus (HCV) infections, excessive alcohol consumption, nonalcoholic fatty liver disease, hemochromatosis, drugs and aflatoxin B1. It is estimated that 70%-90% of patients with HCC have chronic liver disease and cirrhosis, which limits the feasibility of surgical procedures in advanced cases. There are limited treatment options for HCC patients who are ineligible for surgical resection. Locoregional therapies, such as radiofrequency ablation (RFA), transarterial chemoembolization (TACE), transarterial embolization (TAE), or hepatic arterial infusion chemotherapy (HAIC), are primarily recommended, and if one of those fail, then systemic therapy is considered. The 2013 Japan Society of Hepatology HCC Guidelines outlined that the factors influencing treatment decisions should be based on the degree of liver damage (Child-Pugh), presence or absence of extrahepatic spread and macrovascular invasion, the number of tumors, and tumor diameter. Sorafenib has been the standard of care since 2007, when the SHARP trial demonstrated that sorafenib improved median overall survival (OS) compared to placebo in patients who had not received prior systemic therapy (10.7 vs 7.9 months, HR =0.69, P<0.001). In patients from the Asia-Pacific region taking sorafenib, the median improvement in overall survival compared with placebo was 2.3 months (6.5 months vs 4.2 months; HR 0.68; p=0.014). Drug development for hepatocellular carcinoma in the past 10 years has been marked by four failed global phase 3 trials (of sunitinib, brivanib, linifanib, and erlotinib plus sorafenib) that did not show non inferiority. Sorafenib, an oral multikinase inhibitor, has been the only systemic therapy demonstrated to extend overall survibility as a firstline treatment, showing a median improvement of 2.8 months compared with placebo (10.7 months vs. 7.9 months; hazard ratio [HR] 0.69; p\0.001). Inpatients from the Asia-Pacific region taking sorafenib, the median OS (mOS) improvement compared with placebo was 2.3 months (HR 0.68; p = 0.014). The use of other molecularly targeted agents has not demonstrated efficacy via non-inferiority or superiority to sorafenib; thus, until the appearance of lenvatinib, sorafenib has also been widely used as the first-line treatment for HCC patients in Japan. Recently, regorafenib and Nivolumab were approved as a second-line systemic treatment for patients who do not respond to the first-line treatments. Otherwise, best supportive care or participation in clinical trials is recommended in the second-line setting by treatment guidelines. Chemotherapy in combination with sorafenib (doxorubicin), and radioembolization with SIR Spheres Y-90 resin microspheres failed to demonstrate a survival benefit or showed a worse safety profile compared to sorafenib in the first-line setting. Eventually, the PhaseIII non-inferiority REFLECT trial showed that lenvatinib was non-inferior compared to sorafenib.
2. Objectives

   2.1 General objectives:

   To assess and compare the efficacy of Lenvatinib versus Sorafenib in the management of Hepatitis B virus related Hepatocellular Carcinoma.

   2.2 Specific objectives:

   a. To assess and compare the overall survibility of hepatocellular carcinoma patients between the groups of Lenvatinib and Sorafenib. b. To assess and compare the progression free survival outcome between the groups of Lenvatinib and Sorafenib. c. To assess and compare the improvement of liver function tests between the groups of Lenvatinib and Sorafenib. d. To assess and compare the improvement of AFP levels between the groups of Lenvatinib and Sorafenib. e. To assess and compare the improvement of ECOG performance status of the HCC patients between the groups of Lenvatinib and Sorafenib. f. To assess and compare the improvement of Chil-Pugh scores among the HCC patients between the groups of Lenvatinib and Sorafenib. g. To assess and compare the size and number of target lesions by mRECIST criteria among the HCC patients between the groups of Lenvatinib and Sorafenib.
3. Methodology:

The study will be conducted considering the following methodological aspects.

3.1 Study design: An open label randomized clinical control trial study.

3.2 Study duration: From the date of randomization to next 3 months or till death whichever one will be earlier

3.3 Study place: Department of Hepatology, Sir Salimullah Medical College Mitford Hospital

3.4 Study population: Patients diagnosed as advanced Hepatocellular Carcinoma by imaging, cytology or histology with no option of resectibility will be selected for the study.

3.5 Sample size calculation:

"n=" "P1" ("1-P1" )"+P2" ("1-P2" )/("P1" -"P2" )^2 ×〖(Zα+Zβ)〗^2

P1= Proportion of patients developed objective response in one arm (Lenvatinib group) P2= Proportion of patients developed objective response in another arm (Sorafenib group) Zα= Z-value (two tail) at a definite level of significance e.g. 1.96 at 5% level of significance Zβ= Z-value (one tail) at a definite power e.g. 0.84

Here, P1= 40.6% objective response with Lenvatinib (0.406), P2= 12.4% objective response with Sorafenib (0.124), Zα=1.96 and Zβ= 0.8419

n=(0.406(1-0.406)+ 0.124(1-0.124))/〖(0.406-0.124)〗^2 ×〖(1.96+0.84)〗^2 = 34.3 in each group = 35 in each group Total sample number 70 (35 in Lenvatinib group and 35 in Sorafenib group)

3.6 Sampling technique and recruitment of study subjects:

Participants of the study will be recruited via 1:1 randomization from patients admitted in the department of Hepatology, Sir Salimullah Medical College Mitford Hospital and diagnosed as a case of advanced Hepatocellular Carcinoma with no option of resectibility.

3.7 Eligibility criteria:

3.7.1 Inclusion criteria:

1. Patients with Hepatocellular Carcinoma (Diagnosed histologically or cytologically or by imaging criteria with CT or MRI) with no option of resectibility (BCLC stage B or C)
2. Age ≥ 18 years

3.7.2 Exclusion criteria:

1. Patients with very early stage Hepatocellular Carcinoma (BCLC stage 0)
2. Patients with early stage Hepatocellular Carcinoma (BCLC stage A)
3. Patients with terminal stage Hepatocellular Carcinoma (BCLC stage D)
4. Patients with Hepatocellular Carcinoma with obvious invasion to bile duct.
5. Patients who received previous systemic therapy for Hepatocellular Carcinoma.

7. Patients with jaundice (serum bilirubin ≥ 3 mg/dl) 8. Patients with aminotransferases ≥ 5ULN 8. Patients with other co-morbid conditions (COPD, CKD, Heart failure, IHD, pregnancy)

3.7.3 Primary outcome measure:

1. To measure overall survival of the patients from the date of randomization up to 6 months or till death whichever one will be earlier.

3.7.4 Secondary outcome measure:

1. Progression free survival
2. Time to progress
3. Objective response rate
4. Quality of life
5. Assessment of safety

3.8 Outcome measure:

1. Primary endpoint

   a. Overall survibility (From the date of Randomization to next 3 months or till death)
2. Secondary endpoint

   1. Progression free survival
   2. Time to progress
   3. Quality of life measurement (By ECOG performance status)
   4. Liver function tests (By S.Bilirubin, ALT, AST, ALP, Prothrombin time, INR, Serum albumin)
   5. AFP level
   6. Child-turcotte-Pugh score
   7. Tumor assessment by mRECIST criteria.

      3.9 Research instrument

      For collection of primary data about patient a semi-structured questionnaire will be developed based on research objective. Pre-testing of the questionnaire will be done on other patients admitted at the same facility. After the pretesting, amendment of the items and question will be done based on study finding. In the final questionnaire both structured and open questions will be kept.

      A check list will be prepared to compile the data from hospital records, treatment records, outcome of treatment and laboratory investigation reports.

      3.10 Data collection procedure:

      All data will be collected by face-to-face interview of the patients attendant by the researcher at health facility upon their consent and convenience. Socio demographic and personal information will be recorded from patient through interview, with a semi structured pre-tested questionnaire. Information regarding risk factors and risk behavior will be inquired taking effort to minimize the recall bias.

      3.11 Data processing

      Data processing will include data cleaning and quality control check, editing of data, coding of data and data entry into computer. The edited data will be entered on to the template of SPSS® 23.

      3.12 Data analysis

      The edited data will then be entered on to the template of SPSS® 23. For Back ground variables and socio-demographic data descriptive statistics and relative frequency (percentage) will be generated. All data will be presented as mean ± SD. Qualitative data will be analyzed by Chi-square test and quantitative data will be analyzed by student's t-test. Through univariate analysis the base line characteristics and treatment outcome will be compared. The effect of treatment will be identified through Multivariate analysis after adjusting for possible confounders. Relative risk with 95% CI will be generated through binary logistic regression adjusting for all possible confounders. A statistically significant result will be considered when p value < 0.05.

      3.13 Data Presentation

      Data will be presented in the form of table and graphs. Descriptive statistics will be presented with frequency table. Association will be illustrated with cross tables and test statistics will be added in the foot note of the table. Bar and pie charts will be generated to illustrate descriptive statistics.

      4) Ethical considerations

      Approval from the ethical review committee of Sir Salimullah Medical College and Mitford Hospital will be taken prior to commencement of the study. Informed written consent will be taken from the participants after explaining about the details of the study. The participants will be assured that the information acquired will be used for academic purpose. They will be assured of confidentiality, and for the purpose of data analysis no individual data were reported rather de identified data will be preceded for analysis.

      5) Facilities (Resources, Equipments, Chemicals, Subjects etc. required for the study)
      * Principal investigator has full-fledged Department of Hepatology at "Sir Salimullah Medical College Mitford Hospital, Dhaka."
      * "Sir Salimullah Medical College Mitford Hospital, Dhaka" has adequate facilities to carry out all the investigations required for this study.

      "Sir Salimullah Medical College Mitford Hospital, Dhaka" has adequate facility to deal with the adverse effect of the drug under trial as well as management of the subjects of the current study.

      6) Material & methods:

      The study will be conducted in the department of Hepatology, Sir Salimullah Medical College Mitford Hospital. It will be an open label randomized clinical control trial study. Patients admitted in the department of Hepatology, diagnosed as a case of Hepatocellular Carcinoma by imaging or cytopathology or histopathology will be primarily targeted for the study. Initial assessment of each patient will be done by Chil-pugh score, ECOG performance status, Tumor assessment by mRECIST criteria and BCLC staging. According to initial assessment the patients who will fulfill the inclusion criteria (BCLC stage C) will be informed about the study procedure. Patients who will give informed written consent will be randomly assigned 1:1 ratio to receive either Lenvatinib or Sorafenib. Macroscopic portal vein invasion, extrahepatic spread, or both (yes or no), Eastern Cooperative Oncology Group performance status (0 or 1) will be considered as stratification factors. As the study will be open labeled, the treatment will not be masked to the patients or investigators. After randomization there will be two groups; Lenvatinib group (Group A) and Sorafenib group (Group B). Group A patients will receive Cap. Lenvatinib 8 mg/day in two divided doses and group B patients will receive tab. Sorafenib 400 mg/day in two divided doses. Tumor evaluation will be done in each treatment arm in accordance with mRECIST criteria. Liver will be examined with CT or MRI by using a triphasic scanning technique. Patient follow-up and tumor assessment will be done in every 6 weeks interval by liver function tests (S. Bilirubin, ALT, AST, ALP, Prothrombin time, S. Albumin), AFP and imaging (triphasic CT or MRI). Quality of life will be assessed by ECOG performance status on follow-up. Patients will followed up for next 3 months or till death whichever one will be earlier. After 3 months of treatment the two groups (Group A and Group B) will be compared of overall survibility, improvement of patient's clinical and biochemical status, reduction of tumor size as well as the tumor marker.

      7) Statistical Analysis:

      The result of the study will be collected in a separate questionnaire sheet. After collection of data it will be compiled and analyzed using SPSS software version 23.

      References:

1. Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1; 136 (5):359-86. 2. Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31; 391(10127):1301-1314. 3. Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first- line treatment of patients with unresectable hepatocellular carcinoma: A randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24; 391(10126):1163-1173. 4. Snayal AJ, Yoon SK, Lencioni R. The etiology of hepatocellular carcinoma and consequences for treatment. The Oncologist. 2010; 15(4):14-22. 5. Kokudo N, Hasegawa K, Akahane M, Igaki H, Izumi N, Ichida T, Uemoto S, Kaneko S, Kawasaki S, Ku Y, Kudo M, Kubo S, Takayama T, Tateishi R, Fukuda T, Matsui O, Matsuyama Y, Murakami T, Arii S, Okazaki M, Makuuchi M. Evidence-based clinical practice guidelines for hepatocellular carcinoma: The Japan society of Hepatology 2013 update (3rd JHS-HCC guidelines). Hepatol RES. 2015 Jan 27; 45(2): 123-127. 6. Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Häussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med.

2008 Jul 24; 359(4):378-390. 7. Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind,placebo- controlled trial. Lancet Oncol. 2009 Jan; 10(1): 25-34. 8. Cheng AL, Kang YK, Lin DY, Park JW, Kudo M, Qin S, Chung HC, Song X, Xu J, Poggi G, Omata M, Pitman Lowenthal S, Lanzalone S, Yang L, Lechuga MJ, Raymond E. Sunitinib versus sorafenib in advanced hepatocellular cancer: results of a randomized phase III trial. J Clin Oncol. 2013 Nov 10; 31(32): 4067-75. 9. Johnson PJ, Qin S, Park JW, Poon RT, Raoul JL, Philip PA, Hsu CH, Hu TH, Heo J, Xu J, Lu L, Chao Y, Boucher E, Han KH, Paik SW, Robles-Aviña J, Kudo M, Yan L, Sobhonslidsuk A, Komov D, Decaens T, Tak WY, Jeng LB, Liu D, Ezzeddine R, Walters I, Cheng AL. Brivanib versus sorafenib as first-line therapy in patients with unresectable, advanced hepatocellular carcinoma: results from the randomizedphase III BRISK-FL study. J Clin Oncol. 2013 Oct 1; 31(28): 3517-24. 10. Cainap C, Qin S, Huang WT, Chung IJ, Pan H, Cheng Y, Kudo M, Kang YK, Chen PJ, Toh HC, Gorbunova V, Eskens FA, Qian J, McKee MD, Ricker JL, Carlson DM, El-Nowiem S. Linifanib versus sorafenib in patients with advanced hepatocellular carcinoma: results of a randomized phase III trial. J Clin Oncol. 2015 Jan 10; 33(2): 172-79. 11. Zhu AX, Rosmorduc O, Evans TR, Ross PJ, Santoro A, Carrilho FJ, Bruix J, Qin S, Thuluvath PJ, Llovet JM, Leberre MA, Jensen M, Meinhardt G, Kang YK. SEARCH: a phase III, randomized, double-blind, placebo-controlled trial of sorafenib plus erlotinib in patients with advanced hepatocellular carcinoma. J Clin Oncol. 2015 Feb 20;33(6):559-66. 12. Kaneko S, Ikeda K, Matsuzaki Y, Furuse J, Minami H, Okayama Y, Sunaya T, Ito Y, Inuyama L, Okita K. Safety and effectiveness of sorafenib in Japanese patients with hepatocellular carcinoma in daily medical practice: interim analysis of a prospective post marketing all-patient surveillance study. J Gastroenterol. 2016 Oct;51(10):1011- 21. 13. Kudo M, Ikeda M, Takayama T, Numata K, Izumi N, Furuse J, Okusaka T, Kadoya M, Yamashita S, Ito Y, Kokudo N. Safety and efficacy of sorafenib in Japanese patients with hepatocellular carcinoma in clinical practice: a subgroup analysis of GIDEON. J Gastroenterol. 2016 Dec;51(12):1150-60. 14. Bruix J, Qin S, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Breder V, Gerolami R, Masi G, Ross PJ, Song T, Bronowicki JP, Ollivier-Hourmand I, Kudo M, Cheng AL, Llovet JM, Finn RS, LeBerre MA, Baumhauer A, Meinhardt G, Han G; RESORCE Investigators. Regorafenib for patients with hepatocellular carcinoma who progressed on sorafenib treatment (RESORCE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet.

2017 Jan 7;389(10064):55-66. 15. NCCN evidence blocks. Hepatobiliary cancers. NCCN clinical practice guidelines in oncology; 2017. Available from: https://www.nccn.org/professionals/physician_gls/default.aspx. 16. Abou-Alfa GK , Niedzwieski D , Knox JJ , Kaubisch A , Posey J , Kavan BRT , Goel R Murray JJ , Bekaii-Saab TS , Tam VC, Rajdev L , Kelley RK , Siegel A , Balletti J , Harding JJ , Schwartz LH , Goldberg RM , Bertagnolli MM , Venook AP. Phase III randomized study of sorafenib plus doxorubicin versus sorafenib in patients with advanced hepatocellular carcinoma (HCC): CALGB 80802 (Alliance). J Clin Oncol. 2016 Feb 1;34(4):192-192 17. Vilgrain V, Pereira H, Assenat E, Guiu B, Ilonca AD, Pageaux GP, Sibert A, Bouattour M, Lebtahi R, Allaham W, Barraud H, Laurent V, Mathias E, Bronowicki JP, Tasu JP, Perdrisot R, Silvain C, Gerolami R, Mundler O, Seitz JF, Vidal V, Aubé C, Oberti F, Couturier O, Brenot-Rossi I, Raoul JL, Sarran A, Costentin C, Itti E, Luciani A, Adam R, Lewin M, Samuel D, Ronot M, Dinut A, Castera L, Chatellier G; SARAH Trial Group. Efficacy and safety of selective internal radiotherapy with yttrium-90 resin microspheres compared with sorafenib in locally advanced and inoperable hepatocellular carcinoma (SARAH): an open-label randomised controlled Phase 3 trial. Lancet Oncol. 2017 Dec;18(12):1624-1636. 18. Chow PKH, Gandhi M, Tan SB, Khin MW, Khasbazar A, Ong J, Choo SP, Cheow PC, Chotipanich C, Lim K, Lesmana LA, Manuaba TW, Yoong BK, Raj A, Law CS, Cua IHY, Lobo RR, Teh CSC, Kim YH, Jong YW, Han HS, Bae SH, Yoon HK, Lee RC, Hung CF, Peng CY, Liang PC, Bartlett A, Kok KYY, Thng CH, Low AS, Goh ASW, Tay KH, Lo RHG, Goh BKP, Ng DCE, Lekurwale G, Liew WM, Gebski V, Mak KSW, Soo KC; Asia-Pacific Hepatocellular Carcinoma Trials Group. SIRveNIB: selective internal radiation therapy versus sorafenib in Asia-Pacific patients with hepatocellular carcinoma. J Clin Oncol. 2018 Jul 1;36(19):1913-1921. 19. Nicola P, Tiziana P, Lorenza R. Lenvatinib for the treatment of unresectable hepatocellular carcinoma: Evidence to date. Journal of hepatocellular carcinoma.

2019 Jan 31; 6: 31-39. 20. Reig M, Bruix J. Hepatocellular Carcinoma. The Lancet.2018 Mar 31; 391(10127): 1301-1314. 21. Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. AM J Clin Oncol: 1982 Dec; 5(6): 649-655. 22. Lencioni R, Liovet JM. Modified RECIST (mRECIST) Assessment for Hepatocellular Carcinoma. Semin Liver Dis. 2010 Feb; 30 (1): 52-60. 23. Attia KA, Mahassadi AK, Messou E, Kissi YH. Child-Pugh-Turcott versus Meld score for predicting survival in a retrospective cohort of black African cirrhotic patients.

World Gastroenterol. 2008 Jan;14(2): 286-291.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with Hepatocellular Carcinoma (Diagnosed histologically or cytologically or by imaging criteria with CT or MRI) with no option of resectibility (BCLC stage B or C) 2. Age ≥ 18 years

Exclusion Criteria:

- 1. Patients with very early stage Hepatocellular Carcinoma (BCLC stage 0) 2. Patients with early stage Hepatocellular Carcinoma (BCLC stage A) 3. Patients with terminal stage Hepatocellular Carcinoma (BCLC stage D) 4. Patients with Hepatocellular Carcinoma with obvious invasion to bile duct. 5. Patients who received previous systemic therapy for Hepatocellular Carcinoma.

7. Patients with jaundice (serum bilirubin ≥ 3 mg/dl) 8. Patients with aminotransferases ≥ 5ULN 8. Patients with other co-morbid conditions (COPD, CKD, Heart failure, IHD, pregnancy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survivability | From the date of Randomization to next 3 months or till death
  Overall survivability of hepatocellular carcinoma patients will be assessed and compared between two groups (Lenvatinib group vs Sorafenib group)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad S Hossain, MBBS, MD, Principal Investigator — Sir Salimullah Medical College
Locations (2):
- Bangladesh (2):
  - Department of Hepatology, Dhaka
  - Sir Salimullah Medical College, Dhaka

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study and statistical analysis, the study report will be published.
Supporting Information: CSR
Time Frame: January' 2021 - December'2021
Access Criteria: romelssmcmh@gmail.com